CLINICAL TRIAL: NCT02574312
Title: Comparison of Alignment Achieved Using Single-Use Versus Reusable Instrumentation in Total Knee Arthroplasty (TKA): A Prospective, Non-Randomized Multi-center Investigation
Brief Title: ATTUNE Single-Use Instrumentation vs. ATTUNE Reusable Instrumentation in Primary Total Knee Arthroplasty
Acronym: SOLO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10002
Record Dates: First submitted 2015-09-30; First posted 2015-10-12 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis; Post-traumatic Arthritis
Keywords: Mechanical Axis Alignment; Knee Arthroplasty, Total
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TKA with RUI (Active Comparator): 44 Subjects will receive TKA with RUI per their study doctor's standard of care. These 44 subjects will receive the TKA using Reusable instruments (RUI).
  Interventions: Device: ATTUNE TKA with ATTUNE RUI
- TKA with SUI (Experimental): 44 Subjects will receive TKA with SUI per their study doctor's standard of care. These 44 subjects will receive the TKA using Single Use Instruments (SUI).
  Interventions: Device: ATTUNE TKA with ATTUNE SUI

INTERVENTIONS:
Device: ATTUNE TKA with ATTUNE RUI — ATTUNE TKA with ATTUNE RUI
  Other Names: ATTUNE Intuition
  Arms: TKA with RUI
Device: ATTUNE TKA with ATTUNE SUI — ATTUNE TKA with ATTUNE SUI
  Other Names: ATTUNE SOLO
  Arms: TKA with SUI

SUMMARY:
This post-marketing investigation will evaluate the mechanical axis alignment achieved with the ATTUNE Single-Use Instrumentation (SUI) as compared to the mechanical axis alignment achieved with the ATTUNE Reusable Instrumentation (RUI) in primary cemented Total Knee Arthroplasty.

DETAILED DESCRIPTION:
This study is designed as comparative, sequential, non-randomized, multi-center investigation.

Up to four sites will recruit approximately 88 subjects. Each site is expected to implant the ATTUNE primary cemented total knee in approximately 22 subjects. The sequential design requires all ATTUNE TKA with reusable instruments be completed before doing any ATTUNE TKA with single use instruments.

The mechanical axis alignment will be assessed at the 3 month follow-up by independent radiographic review.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with severely painful and/or severely disabling Non-inflammatory Degenerative Joint Disease (NIDJD) resulting from osteoarthritis (OA) or post-traumatic arthritis.
2. Subject is male or female and between the ages of 22 and 80 years old, inclusive.
3. Subject requires a primary total knee replacement and is considered by the Investigator to be suitable for the specific knee prosthesis identified in the protocol.
4. Subject, who, in the opinion of the Investigator, is suitable for implantation using either RUI or SUI instrumentation.
5. Subject is able to speak and read English to facilitate comprehension of the Informed Consent Document.
6. Subject has given voluntary, written informed consent to participate in this clinical investigation and has authorized the transfer of his/her information to DePuy Synthes Joint Reconstruction.
7. Subject, in the opinion of the Investigator, is able to understand this clinical investigation and is willing and able to perform all study procedures and follow-up visits and co-operate with investigational procedures.

Exclusion Criteria:

1. The Subject has, in the opinion of the Investigator, a severe deformity that will hinder achieving a mechanical axis alignment target of 0° ± 3°.
2. The Subject has, in the opinion of the Investigator, an existing condition that would compromise their participation and follow-up in this study.
3. The Subject has, in the opinion of the Investigator, a flexion deformity that will not allow for 0° extension postoperatively.
4. The Subject is a woman who is pregnant or lactating.
5. The Subject, in the opinion of the Investigator, is a drug or alcohol abuser (in the last 5 years) or has a psychological disorder that could affect follow-up care or treatment outcomes.
6. The Subject has participated in a clinical investigation with an investigational product in the last 3 months.
7. The Subject is currently involved in any personal injury litigation, medical-legal or worker's compensations claims.
8. The Subject has previous prosthetic knee replacement (any type including unicompartmental, total knee arthroplasty, patellofemoral arthroplasty or ipsilateral UTO/HTO) of the affected knee or a previous patellectomy.
9. The Subject presents with ankylosis of the hip joint on the side to be treated.
10. The Subject had a contralateral TKA and that knee was previously entered into the study.
11. The Subject requires simultaneous bilateral total knee replacements.
12. Any case in which Computer-Assisted Surgery (CAS) or TruMatch (or any other type of Custom Patient Instruments) is to be used, or any additional instrumentation are to be used for bone resections that are not provided as part of the ATTUNE RUI or SUI Instrument kits.
13. The Subject requires a device not specified in the protocol or the surgeon determines that the ATTUNE Knee System is not a suitable treatment.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Verdonna Huey, MS,BSN,CCRP, Study Director — DePuy Synthes
Locations (4):
- United States (2):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
- United Kingdom (2):
  - Spire Liverpool Hospital, Liverpool
  - Clifton Park Hospital, York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient was operated on 16 November 2015 and recruitment lasted for 37 months with the last patient operated on 19 December 2018.
Pre-assignment Details: Consent was taken for 102 knees, 14 subjects were deemed ineligible for the study. This left 88 subjects in the safety population that could be randomised for the study.
Groups:
- RUI (Reuseable Instrumentation): Patients were operated on using Reusable TKA Instrumentation
- SUI (Single-Use Instrumentation): Patients were operated on using Single-Use TKA Instrumentation
Period: Pre-Operative
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0
Period: 3 Months Follow-up
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Started | 44 | 44
Completed | 43 (One subject withdrew consent) | 44
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects who received the study device.
Groups:
- Total: Total of all reporting groups
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation) | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (6.89) | 69.3 (7.98) | 67.9 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 24 | 18 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 22 | 22 | 44
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 22 | 22 | 44
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Difference in Absolute Mechanical Axis Alignment Angle Between Subjects Operated on With RUI and SUI TKA Instrumentation
Time Frame: 3 Months Post Surgery
Population: All patients with readable radiographs who were enrolled without major protocol violations
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Radiographs
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 34 | 41
Number analyzed (Radiographs) | 34 | 41
Degrees | 2.55 (2.44) | 2.97 (2.33)
Statistical Analysis 1: Comparison: RUI (Reuseable Instrumentation) vs SUI (Single-Use Instrumentation); Test type: Non-Inferiority — Non-Inferiority Analysis of absolute value of mechanical axis alignment with NI margin of 1.5 degrees, using a 1-sided T-test with alpha of 0.05. Anticipated power was 95%; p = 0.028, t-test, 1 sided

2. Secondary Outcome: Femoral Component Varus Valgus Angle Between Subjects Operated on With RUI and SUI TKA Instrumentation
Time Frame: 3 Months Post Surgery
Population: All patients with readable radiographs who were enrolled without major protocol violations
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Radiographs
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 34 | 41
Number analyzed (Radiographs) | 34 | 41
Degrees | 94.9 (2.10) | 95.8 (2.40)

3. Secondary Outcome: Tibial Component Varus Valgus Angle Between Subjects Operated on With RUI and SUI TKA Instrumentation
Time Frame: 3 Months Post Surgery
Population: All patients with readable radiographs who were enrolled without major protocol violations
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Radiographs
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 34 | 41
Number analyzed (Radiographs) | 34 | 41
Degrees | 88.4 (2.18) | 88.7 (2.23)

4. Secondary Outcome: Femoral Component Flexion Angle Between Subjects Operated on With RUI and SUI Instrumentation
Time Frame: 3 Months Post Surgery
Population: All patients with readable radiographs who were enrolled without major protocol violations
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Radiographs
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 34 | 41
Number analyzed (Radiographs) | 34 | 41
Degrees | 6.21 (2.70) | 7.91 (3.20)

5. Secondary Outcome: Posterior Tibial Slope Between Subjects Operated on With RUI and SUI Instrumentation
Time Frame: 3 Months Post Surgery
Population: All patients with readable radiographs who were enrolled without major protocol violations
Measure: Mean (Standard Deviation); unit: Degrees
Units Other Than Participants: Radiographs
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 34 | 41
Number analyzed (Radiographs) | 34 | 41
Degrees | 1.04 (2.49) | 0.78 (2.70)

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Time Frame: 3 Months Post Surgery
Population: All subjects who received the study device
Measure: Number; unit: Participants
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
Number analyzed (Participants) | 44 | 44
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All participants had reached the 3 month follow-up visit at the time of uploading adverse events.
Description: Final assessment of adverse events were classified by system organ class in lieu of specific adverse event terms.
Arm/Group | RUI (Reuseable Instrumentation) | SUI (Single-Use Instrumentation)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/44 | 0/44
Other Adverse Events (participants affected / at risk) | 5/44 | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RUI (Reuseable Instrumentation) (N=44) | SUI (Single-Use Instrumentation) (N=44)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RUI (Reuseable Instrumentation) (N=44) | SUI (Single-Use Instrumentation) (N=44)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Vascular (Vascular disorders) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 1 (1) | 1 (1)
Immune System Disorder (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
DePuy reserves the right to review the contents of publications in advance.The PI may freely disclose the trial results only after DePuy has been given the opportunity of reviewing the proposed results communications at least 30 days prior to the intended release.DePuy will advise the PI of any perceived errors,omissions or corrections but PI will retain final editorial control. In case of disagreement, DePuy and PI will make every effort to meet in order to discuss and resolve any issues.

DOCUMENTS (2):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT02574312/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/12/NCT02574312/SAP_001.pdf